CLINICAL TRIAL: NCT04597632
Title: A 56-week Phase IIIb/IV, Open-label, One-arm Extension Study to Assess the Efficacy and Safety of Brolucizumab 6 mg in a Treat-to-Control Regimen With Maximum Treatment Intervals up to 20 Weeks for the Treatment of Patients With Neovascular Age-related Macular Degeneration Who Have Completed the CRTH258A2303 (TALON) Study
Brief Title: An Extension Study Assessing the Efficacy and Safety of Brolucizumab in a Treat-to-Control Regimen in Patients With Neovascular Age-related Macular Degeneration Who Have Completed the CRTH258A2303 (TALON) Study
Acronym: TALON Ext
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRTH258A2303E1; 2020-002349-40 (EudraCT Number)
Record Dates: First submitted 2020-10-01; First posted 2020-10-22 (Actual); Results first posted 2024-04-04 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Neovascular Age-related Macular Degeneration
Keywords: neovascular age-related macular degeneration; wet age-related macular degeneration; wet AMD; choroidal neovascularization; individualized treatment; anti-VEGF; Macular degeneration; age-related macular degeneration (ARMD); vision loss; macula damage; retina damage; dry macular degeneration; wet macular degeneration; Subfoveal choroidal neovascularization (CNV) secondary to age-related macular degeneration
MeSH Terms: conditions — Choroidal Neovascularization; Macular Degeneration; Vision Disorders; Geographic Atrophy; Wet Macular Degeneration | interventions — brolucizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- brolucizumab 6 mg (Experimental): Participants received brolucizumab 6 mg/0.05 mL solution by intravitreal injection in a Treat-to-Control regimen with injection intervals from 4 up to 20 weeks. Intervals could have changed in steps of 4 weeks at a time per investigators' decisions determined by the disease activity.
  Interventions: Drug: brolucizumab

INTERVENTIONS:
Drug: brolucizumab — brolucizumab 6 mg/0.05 mL solution for intravitreal injection
  Other Names: RTH258

SUMMARY:
The purpose of this extension study was to evaluate the efficacy and safety of brolucizumab used in a Treat-to-Control-regimen for treatment of patients with neovascular age-related macular degeneration who have completed the CRTH258A2303 (TALON) study. The main objective was to assess brolucizumab's potential for long durability up to 20 weeks.

All eligible participants were treated with brolucizumab regardless of their treatment in the TALON study.

The study period was 56 weeks including post-treatment follow-up.

DETAILED DESCRIPTION:
This was a 56-week, open-label, one-arm extension study in subjects who had completed the CRTH258A2303 (TALON) (NCT04005352) study, referred to as the core study in this document. Subjects who provided written informed consent and met all the inclusion and none of the exclusion criteria were enrolled into this extension study to receive brolucizumab 6 mg in a treat-to-control (TtC) regimen, irrespective of the treatment received in the core study.

The maximum study duration for a subject was 56 weeks, including post-treatment follow-up.

There were two periods in this study:

* Treat-to-Control treatment period: from Baseline (Day 1) to Week 52
* Post-treatment follow-up period: from Week 52 to Week 56.

All participants were treated with brolucizumab regardless of their treatment in the TALON study (brolucizumab or aflibercept).

Treatment intervals were then extended by 4 weeks at a time based on the investigator's judgment of visual and/or anatomic outcomes. The treatment intervals were to have been 4 weeks at a time if disease activity recurs.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Successfully completed TALON core study at week 64 (End of Study)

Exclusion Criteria:

1. Medical condition or personal circumstance which precludes study participation or compliance with study procedures, as assessed by the Investigator
2. Discontinued study treatment in the core study
3. Anti-VEGF treatment is futile in the study eye, in the Investigator's opinion.
4. Pregnant or nursing (lactating) women
5. Women of child-bearing potential not using highly effective methods of contraception

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2020-12-16 (Actual); Primary Completion 2023-03-28 (Actual); Study Completion 2023-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (55):
- United States (5):
  - Novartis Investigative Site, Huntington Beach, California
  - Novartis Investigative Site, Fort Lauderdale, Florida
  - Novartis Investigative Site, Indianapolis, Indiana
  - Novartis Investigative Site, Minneapolis, Minnesota
  - Novartis Investigative Site, Germantown, Tennessee
- Australia (7):
  - Novartis Investigative Site, Albury, New South Wales
  - Novartis Investigative Site, Hurstville, New South Wales
  - Novartis Investigative Site, Parramatta, New South Wales
  - Novartis Investigative Site, Sydney, New South Wales
  - Novartis Investigative Site, Glen Waverley, Victoria
  - Novartis Investigative Site, Rowville, Victoria
  - Novartis Investigative Site, Nedlands, Western Australia
- Novartis Investigative Site, Hasselt, Belgium
- Czechia (2):
  - Novartis Investigative Site, Hradec Králové, CZE
  - Novartis Investigative Site, Prague
- France (9):
  - Novartis Investigative Site, Saint-Cyr-sur-Loire, Indre Et Loire
  - Novartis Investigative Site, Lyon, Rhone
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Créteil
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Montauban
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Rueil-Malmaison
- Germany (3):
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Mainz
- Israel (3):
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Ramat Gan
  - Novartis Investigative Site, Ẕerifin
- Novartis Investigative Site, Perugia, PG, Italy
- Malaysia (3):
  - Novartis Investigative Site, Malacca, Melaka Malaysia
  - Novartis Investigative Site, Batu Caves, Selangor
  - Novartis Investigative Site, Shah Alam, Selangor
- Netherlands (2):
  - Novartis Investigative Site, 's-Hertogenbosch
  - Novartis Investigative Site, Nijmegen
- Portugal (2):
  - Novartis Investigative Site, Porto
  - Novartis Investigative Site, Vila Franca de Xira
- South Korea (5):
  - Novartis Investigative Site, Bundang Gu, Gyeonggi-do
  - Novartis Investigative Site, Seoul, Seocho Gu
  - Novartis Investigative Site, Busan
  - Novartis Investigative Site, Daegu
  - Novartis Investigative Site, Seoul
- Spain (7):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Sant Cugat del Vallès, Catalonia
  - Novartis Investigative Site, Pamplona, Navarre
  - Novartis Investigative Site, Burjassot, Valencia
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Córdoba
  - Novartis Investigative Site, Zaragoza
- Sweden (2):
  - Novartis Investigative Site, Örebro
  - Novartis Investigative Site, Västerås
- Novartis Investigative Site, Binningen, Switzerland
- Taiwan (2):
  - Novartis Investigative Site, Taipei
  - Novartis Investigative Site, Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on https://www.clinicalstudydatarequest.com/.
URL: https://www.clinicalstudydatarequest.com/

REFERENCES:
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1913

RESULTS

PARTICIPANT FLOW:
Groups:
- Brolucizumab 6 mg (Extension Study Total): Participants received brolucizumab 6 mg/0.05 mL solution by intravitreal injection in a Treat-to-Control regimen with injection intervals from 4 up to 20 weeks. Intervals could have changed in steps of 4 weeks at a time per investigators' decisions determined by the disease activity.
Period: Overall Study
Arm/Group | Brolucizumab 6 mg (Extension Study Total)
Started | 248
Completed | 231
Not Completed | 17
Not completed — Withdrawal by Subject | 10
Not completed — Lost to Follow-up | 1
Not completed — Death | 1
Not completed — Adverse Event | 5

BASELINE CHARACTERISTICS:
Population: Full Analysis Set composed of all subjects who received at least one dose of study treatment in the extension study.
Arm/Group | Brolucizumab 6 mg (Extension Study Total)
Number analyzed (Participants) | 248
Age, Continuous [Mean (Standard Deviation); unit: Years] | 75.9 (7.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 129
  Male | 119
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23
  Not Hispanic or Latino | 219
  Unknown or Not Reported | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 61
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 187
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Duration of the Last Interval With no Disease Activity up to Week 56 - Study Eye
Description: Number of subjects in every 4 weeks (q4w), every 8 weeks (q8w), every 12 weeks (q12w) and every 20 weeks (q20w) intervals at last interval with no disease activity up to Week 56. Last interval with no disease activity (number of weeks): Number of subjects at 20/16/12/8/4-weeks intervals up to Week 56 for the study eye in the extension study
Time Frame: Up to Week 56
Population: Full Analyses Set. Subjects with at least two injections in the extension study
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg
Number analyzed (Participants) | 237
Participants
  20 weeks | 68
  16 weeks | 59
  12 weeks | 47
  8 weeks | 49
  4 weeks | 14

2. Primary Outcome: Average Change in BCVA From Baseline to Week 52 and Week 56 for the Study Eye
Description: Best-Corrected Visual Acuity (BCVA) was assessed using Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity testing charts. Visual Function of the study eye was assessed using the ETDRS protocol. Min and max possible scores are 0-100 respectively. A higher score represents better visual functioning.
  The average change in BCVA from Baseline of the extension study at Week 52 and Week 56 was estimated by an analysis of variance (ANOVA) with baseline age categories, baseline BCVA categories and treatment arm in the core study included as fixed effects. Last observation carried forward (LOCF) was used to impute missing BCVA values.
Time Frame: Extension study baseline, average of Week 52 and Week 56
Population: Full Analyses Set - Last Observation Carried Forward. Participants were analyzed according to the originally assigned treatment arm in the core study (CRTH258A2303, NCT04005352).
Measure: Mean (Standard Deviation); unit: Letters read
Groups:
- Brolucizumab 6 mg (Core Study): Patients who received brolucizumab 6 mg in the core study and continued with the same treatment in the extension study
- Aflibercept 2 mg (Core Study): Patients who received aflibercept 2 mg in the core study and switched to brolucizumab 6 mg in the extension study
Arm/Group | Brolucizumab 6 mg (Core Study) | Aflibercept 2 mg (Core Study) | Brolucizumab 6 mg (Extension Study Total)
Number analyzed (Participants) | 135 | 113 | 248
Letters read | -1.8 (8.29) | -2.9 (7.33) | -2.3 (7.88)

3. Secondary Outcome: Average Change in Central Subfield Thickness (CSFT) From Baseline to Week 52 and Week 56 - Study Eye
Description: Central Subfield Thickness (μm): Analysis of Variance (ANOVA) results for the average change from extension study Baseline at Week 52 and Week 56 for the study eye in the extension study by core study treatment arm.
  Central Subfield Thickness was assessed by Spectral domain optical coherence tomography (SD-OCT) from the central reading center.
Time Frame: Extension study baseline, average of Week 52 and Week 56
Population: Participants in the Full Analysis Set with a valid measurement for the outcome measure. Participants were analyzed according to the originally assigned treatment arm in the core study (CRTH258A2303, NCT04005352).
Measure: Mean (Standard Deviation); unit: μm
Arm/Group | Brolucizumab 6 mg (Core Study) | Aflibercept 2 mg (Core Study) | Brolucizumab 6 mg (Extension Study Total)
Number analyzed (Participants) | 105 | 89 | 194
μm | 5.9 (24.43) | -14.1 (60.67) | -3.3 (45.83)

4. Secondary Outcome: Number (%) of Subjects With Presence of IRF and/or SRF, and Sub-RPE Fluid in the Study Eye at Week 52 and Week 56 Overall and by Core Study Treatment Arm
Description: Intraretinal Fluid (IRF) and Subretinal Fluid (SRF) status in the central subfield as assessed by Spectral Domain Ocular Coherence Tomography (SD-OCT): Number (%) of subjects with presence of IRF and/or SRF, and sub-Retinal Pigment Epithelium (RPE) fluid in the study eye at Week 52 and Week 56 overall and by core study treatment arm
Time Frame: Weeks 52 and 56
Population: Full Analyses Set - for subjects with a valid measurement
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg (Core Study) | Aflibercept 2 mg (Core Study) | Brolucizumab 6 mg (Extension Study Total)
Number analyzed (Participants) | 106 | 94 | 200
Participants
  Week 52 IRF assessment - Present (n=103,90,193): number analyzed (Participants) | 103 | 90 | 193
  Week 52 IRF assessment - Present (n=103,90,193) | 10 | 14 | 24
  Week 52 IRF assessment - Absent (n=103,90,193): number analyzed (Participants) | 103 | 90 | 193
  Week 52 IRF assessment - Absent (n=103,90,193) | 93 | 76 | 169
  Week 52 SRF assessment - Present (n=103,90,193): number analyzed (Participants) | 103 | 90 | 193
  Week 52 SRF assessment - Present (n=103,90,193) | 14 | 9 | 23
  Week 52 SRF assessment - Absent (n=103,90,193): number analyzed (Participants) | 103 | 90 | 193
  Week 52 SRF assessment - Absent (n=103,90,193) | 89 | 81 | 170
  Week 52 Sub-RPE fluid - Present (n=103,90,193): number analyzed (Participants) | 103 | 90 | 193
  Week 52 Sub-RPE fluid - Present (n=103,90,193) | 52 | 44 | 96
  Week 52 Sub-RPE fluid - Absent (n=103,90,193): number analyzed (Participants) | 103 | 90 | 193
  Week 52 Sub-RPE fluid - Absent (n=103,90,193) | 51 | 46 | 97
  Week 52 IRF and/or SRF - Present (n=103,90,193): number analyzed (Participants) | 103 | 90 | 193
  Week 52 IRF and/or SRF - Present (n=103,90,193) | 23 | 22 | 45
  Week 52 IRF and/or SRF - Absent (n=103,90,193): number analyzed (Participants) | 103 | 90 | 193
  Week 52 IRF and/or SRF - Absent (n=103,90,193) | 102 | 89 | 191
  Week 52 IRF and SRF - Present (n=103,90,193): number analyzed (Participants) | 103 | 90 | 193
  Week 52 IRF and SRF - Present (n=103,90,193) | 1 | 1 | 2
  Week 52 IRF and SRF - Absent (n=103,90,193): number analyzed (Participants) | 103 | 90 | 193
  Week 52 IRF and SRF - Absent (n=103,90,193) | 80 | 68 | 148
  Week 56 IRF assessment - Present | 13 | 12 | 25
  Week 56 IRF assessment - Absent | 93 | 82 | 175
  Week 56 SRF assessment - Present | 11 | 7 | 18
  Week 56 SRF assessment - Absent | 95 | 87 | 182
  Week 56 Sub-RPE fluid - Present | 51 | 49 | 100
  Week 56 Sub-RPE fluid - Absent | 55 | 45 | 100
  Week 56 IRF and/or SRF - Present | 23 | 17 | 40
  Week 56 IRF and/or SRF - Absent | 105 | 92 | 197
  Week 56 IRF and SRF - Present | 1 | 2 | 3
  Week 56 IRF and SRF - Absent | 83 | 77 | 160

5. Secondary Outcome: Last Interval With no Disease Activity (Number of Weeks): Number (%) of Subjects at 20/16/12/8/4-weeks Intervals up to Week 56 for the Study Eye in the Extension Study by Core Study Randomized Treatment Arm
Description: Duration of the last interval with no disease activity up to Week 52 by core study treatment arm.
Time Frame: up to Week 56
Population: Full Analyses Set - for Subjects with at least two injections in the extension study
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg (Core Study) | Aflibercept 2 mg (Core Study)
Number analyzed (Participants) | 130 | 107
Participants
  20 Weeks | 49 | 19
  16 Weeks | 29 | 30
  12 Weeks | 21 | 26
  8 Weeks | 23 | 26
  4 Weeks | 8 | 6

6. Secondary Outcome: Maximal Interval With no Disease Activity (Number of Weeks): Number (%) of Subjects at 20/16/12/8/4-weeks Intervals up to Week 56 for the Study Eye in the Extension Study
Description: Duration of the maximal intervals with no disease activity up to Week 52 by core study treatment arm.
Time Frame: up to Week 56
Population: Full Analyses Set - for Subjects with at least two injections in the extension study
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg (Core Study) | Aflibercept 2 mg (Core Study)
Number analyzed (Participants) | 130 | 107
Participants
  20 Weeks | 54 | 20
  16 Weeks | 28 | 31
  12 Weeks | 23 | 34
  8 Weeks | 22 | 18
  4 Weeks | 3 | 4

7. Secondary Outcome: Number (%) of Subjects With Change in Duration of Last Interval With no Disease Activity Between Baseline of the Extension Study and Week 56 by Core Study Treatment Arm
Description: Change in last interval with no disease activity
Time Frame: Extension study baseline, up to Week 56
Population: Full Analyses Set - for Subjects with at least two injections in the extension study
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg (Core Study) | Aflibercept 2 mg (Core Study)
Number analyzed (Participants) | 130 | 107
Participants
  16 Weeks | 0 | 2
  12 Weeks | 8 | 5
  8 Weeks | 21 | 32
  4 Weeks | 49 | 28
  0 Weeks | 41 | 31
  - 4 Weeks | 8 | 7
  -8 Weeks | 2 | 2
  -12 Weeks | 1 | 0

8. Secondary Outcome: Treatment-emergent Ocular Adverse Events (Greater Than or Equal to 1.0%) by Preferred Term for the Study Eye
Description: An adverse event (AE) is any untoward medical occurrence (e.g. any unfavorable and unintended sign [including abnormal laboratory findings], symptom or disease) in a clinical investigation participant after providing written informed consent for participation in the study.
Time Frame: Adverse events are reported from the first dose of study-drug until the end of treatment at week 52, plus 4 weeks safety follow-up, for a maximum timeframe of approximately 56 weeks.
Population: Full Analyses Set
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg
Number analyzed (Participants) | 248
Participants
  Number of subjects with at least one AE | 63
  Cataract | 9
  Eye pain | 6
  Visual acuity reduced | 6
  Intraocular pressure increased | 5
  Retinal haemorrhage | 4
  Ocular discomfort | 3
  Vitreous floaters | 3

9. Secondary Outcome: Treatment-emergent Non-ocular Adverse Events (Greater Than or Equal to 2%) by Preferred Term
Description: as for outcome 8
Time Frame: as for outcome 8
Population: Full Analyses Set
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg
Number analyzed (Participants) | 248
Participants
  Number of subjects with at least one AE | 82
  COVID-19 | 10
  Nasopharyngitis | 8
  Fall | 7
  Basal cell carcinoma | 5

10. Post Hoc Outcome: All Collected Deaths
Description: On treatment death monitoring occurred after the first dose of study drug in the extension study until 30 days after the last administration of study drug for a maximum timeframe of approximately 56 weeks. Post-treatment death monitoring occurred greater than 30 days after the last administration of study drug.
Time Frame: On-treatment death reporting - from first dose until 30 days after last dose for a maximum timeframe of approximately 56 weeks. Post-treatment death reporting - greater than 30 days after the last dose of study drug.
Population: Full Analyses Set
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg
Number analyzed (Participants) | 248
Participants
  On-treatment Deaths | 0
  Post-treatment Deaths | 1
  Total Deaths | 1

ADVERSE EVENTS:
Time Frame: Adverse events are reported from the first dose of study-drug until the end of treatment at week 52, plus 4 weeks safety follow-up, for a maximum timeframe of approximately 56 weeks.
Description: Adverse events and the death are reported in the Full Analysis Set that includes all participants who received at least one dose of study treatment in the extension study.
Groups:
- Brolucizumab 6mg: Brolucizumab 6mg
Arm/Group | Brolucizumab 6mg
All-Cause Mortality (participants affected / at risk) | 1/248
Serious Adverse Events (participants affected / at risk) | 26/248
Other Adverse Events (participants affected / at risk) | 58/248
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brolucizumab 6mg (N=248)
Atrial fibrillation (Cardiac disorders) | 2
Retinal detachment - Fellow eye (Eye disorders) | 1
Retinal occlusive vasculitis - Study eye (Eye disorders) | 1
Uveitis - Study eye (Eye disorders) | 1
Vitreal cells - Fellow eye (Eye disorders) | 1
Vitreal cells - Study eye (Eye disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Pneumonia (Infections and infestations) | 1
Pyelonephritis acute (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Whipple's disease (Infections and infestations) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 2
Lower limb fracture (Injury, poisoning and procedural complications) | 1
Meniscus injury (Injury, poisoning and procedural complications) | 1
Procedural vomiting (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Chondropathy (Musculoskeletal and connective tissue disorders) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ischaemic stroke (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Delirium (Psychiatric disorders) | 1
Calculus urinary (Renal and urinary disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Brolucizumab 6mg (N=248)
Cataract - Fellow eye (Eye disorders) | 7
Cataract - Study eye (Eye disorders) | 9
Eye pain - Study eye (Eye disorders) | 6
Neovascular age-related macular degeneration - Fellow eye (Eye disorders) | 10
Visual acuity reduced - Study eye (Eye disorders) | 6
COVID-19 (Infections and infestations) | 10
Nasopharyngitis (Infections and infestations) | 8
Fall (Injury, poisoning and procedural complications) | 7
Intraocular pressure increased - Study eye (Investigations) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-10-20): https://cdn.clinicaltrials.gov/large-docs/32/NCT04597632/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-05): https://cdn.clinicaltrials.gov/large-docs/32/NCT04597632/SAP_001.pdf